CLINICAL TRIAL: NCT07127822
Title: A Randomized, Controlled, Non Inferiority Phase II Clinical Study Comparing Iparomlimab and Tuvonralimab With Standard Chemotherapy Combined With PD-1/PD-L1 Monoclonal Antibody as First-line Treatment for MSI-H/dMMR Recurrent/Metastatic Gastric Cancer
Brief Title: Assessing Iparomlimab and Tuvonralimab in Recurrent or Metastatic MSI-H/dMMR Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Qilu Pharmaceutical Group Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUCH MSI-H GC 1st
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Gastric / Gastroesophageal Junction Adenocarcinoma; MSI-H Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): iparomlimab and tuvonralimab
  Interventions: Drug: Iparomlimab and Tuvonralimab
- Control arm (Active Comparator): standard first-line chemotherapy（FOLFOX/XELOX/SOX） combined with PD-1/PD-L1 antibody
  Interventions: Drug: First line chemotherapy plus PD-1/PD-L1 antibody

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab — Iparomlimab and tuvonralimab for experimental arm
  Arms: Experimental arm
Drug: First line chemotherapy plus PD-1/PD-L1 antibody — standard first-line chemotherapy（FOLFOX/XELOX/SOX）combined with PD-1/PD-L1 antibody for control arm
  Arms: Control arm

SUMMARY:
A randomized controlled phase II study exploring first-line treatment options for recurrent/metastatic MSI-H gastric cancer

DETAILED DESCRIPTION:
This is a randomized controlled, non-inferiority design phase II study in the first-line treatment of recurrent/metastatic MSI-H gastric cancer, using iparomlimab and tuvonralimab and standard first-line chemotherapy combined with PD-1/PD-L1 antibody in two cohorts, respectively,

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily willing to participate in the study and sign the written informed consent form 2. Age ≥18 years male or female . 3. Expected survival time ≥ 3 months 4. Patients with unresectable locally advanced, recurrent, or metastatic gastric/gastroesophageal junction adenocarcinoma diagnosed by histological or cytological examination: 5. Confirmed by PCR or next-generation sequencing(NGS) as microsatellite instability-high(MSI-H) . Patients with mismatch repair defecient identified by immunohistochemistry need to undergo PCR/NGS verification as MSI-H before treatment 6. Patients should not receive systematic anti-tumor treatment before, and for those who have received induction chemotherapy, concurrent radiochemotherapy, or neoadjuvant/adjuvant chemotherapy for curative purposes, the recurrence time must be at least 6 months from the end of the last treatment; 7. Agree to provide archived tumor tissue specimens or fresh tissue samples of primary or metastatic lesions within 3 years; If the patinet is unable to provide tumor tissue samples, they can be enrolled after evaluation by the researcher, provided that they meet other inclusion and exclusion criteria; 8. Patients must have at least one measurable lesion defined by RECIST 1.1. 9. European Cooperative Oncology Group (ECOG) ≤1 10. No severe cardiac dysfunction, left ventricular ejection fraction ≥ 50%; 11. Patients must meet the following criteria at screening and before preconditioning (baseline). If any laboratory test result is abnormal referring to the following criteria,

1. Hematology: neutrophils (NE) ≥1.5×109 per liter, , platelets (PLT) ≥100×109per liter and hemoglobin (Hb) ≥8.0 g/dL.
2. Blood chemistry: creatinine clearance ≥50 mL/min, Creatinine (Cr) ≤ 1.5 × ULN, alanine aminotransferase (ALT) ≤2.5×ULN（Gilbert syndrome or liver metastasis subjects ≤ 5 × ULN）, aspartate aminotransferase (AST) ≤2.5×ULN（Gilbert syndrome or liver metastasis subjects ≤ 5 × ULN）, total bilirubin (TB) ≤1.5×ULN（Gilbert syndrome or liver metastasis subjects ≤ 3 × ULN）,
3. International normalized ratio (INR) ≤ 1.5, and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; 12. Urinary protein ≤ 2+or < 1000mg/24h; 13. Women of childbearing potential must have negative serum pregnancy test result at screening and before preconditioning and agree to use an effective and reliable contraceptive method for at least 1 year after the last study treatment. Te acceptable methods include bilateral tubal ligation/bilateral salpingectomy or bilateral tubal occlusion; any approved oral, injection or implantation of hormone; or barrier contraceptive method: condoms containing spermicidal .

Exclusion Criteria:

1. Pregnant or lactating women.
2. Previous use of PD-1/PD-L1 monoclonal antibodies, CTLA-4 monoclonal antibodies, or monoclonal and bispecific drugs containing the aforementioned targets;
3. Existence of any active autoimmune disease or history of autoimmune disease (such as but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; asthma in which subjects require bronchodilators for medical intervention cannot be included); However, the following diseases are allowed to be included: vitiligo, psoriasis, alopecia without systemic treatment, well controlled type I diabetes, hypothyroidism with normal thyroid function after replacement treatment;
4. Patients who require immunosuppressive therapy, systemic or absorbable local hormone therapy to achieve immunosuppressive goals (calculated as prednisone, dose>10mg/day or other therapeutic hormones) and continue to use it within 2 weeks of the first administration;
5. Patients with uncontrolled pleural effusion, pericardial effusion, or ascites that require repeated drainage;
6. Patients with uncontrollable symptoms of brain metastasis, spinal cord compression, malignant meningitis, or brain or pia mater diseases detected by CT or MRI examination during screening within 4 weeks before the first administration
7. Patients who have received non systematic anti-tumor therapy within 3 weeks prior to the start of treatment, including but not limited to surgery, radiation therapy, interventional therapy, and anti-tumor traditional Chinese medicine treatment (based on the indications in the Chinese medicine instructions, and may also be enrolled after a 2-week washout period). Patients whose adverse events caused by previous treatment (excluding hair loss) have not recovered to ≤ CTCAE grade 2 are not within the above range;
8. Patients with any severe and/or uncontrolled illnesses, including:

1) Patients with poor blood pressure control (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 90 mmHg) 2) Patients who experience unstable angina, myocardial infarction, ≥ grade 2 congestive heart failure, or arrhythmia requiring treatment within 6 months of initial administration (including QTc ≥ 480ms); 3) Active or uncontrolled severe infection (≥ CTCAE grade 2 infection); 4) A history of clinically significant liver disease, including viral hepatitis, known as a carrier of hepatitis B virus (HBV), must exclude active HBV infection, i.e. HBV DNA positive (>2000 IU/mL); Known hepatitis C virus infection (HCV) and HCV RNA positivity (>1 × 103 copies/mL), or other decompensated liver diseases or chronic hepatitis requiring antiviral therapy; 5) HIV test positive 6) Poor control of diabetes (fasting blood glucose ≥ CTCAE level 2); 9. Patients who have experienced severe infections (CTCAE>grade 2) within the first 4 weeks of randomization, such as severe pneumonia, bacteremia, sepsis, tuberculosis, etc; Indications of pulmonary infection or active pulmonary inflammation within the first 2 weeks of randomization; 10. Patients with a history of allergies to recombinant humanized antibodies who are allergic to any excipient components of the drug; 11. History of autologous or allogeneic stem cell transplantation; 12. Patients with a history of serious neurological or psychiatric disorders, including but not limited to: dementia, depression, epileptic seizures, bipolar disorder, etc; 13. Patients diagnosed as active malignant tumor within the first 3 years of randomization, except for the following cases: radical skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, breast carcinoma in situ and/or radical resection of carcinoma in situ, which the researchers think can be included; 14. Patients who plan to receive live vaccines within 28 days prior to randomization; 15. Researchers evaluate situations where participation in this clinical trial is inappropriate due to complications or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Antitumor efficacy-Objective response rate (ORR) | 2 years
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%).

SECONDARY OUTCOMES:
Antitumor efficacy-Progression-free survival (PFS) | 2 years
  The period from the day of randomization to the first recorded tumor progression (whether treated or not) or death of any cause, which occurs first.
Antitumor efficacy-Overall survival (OS) | 2 yeas
  The period from the day of randomization to any cause of death
Treatment related AEs | 2 years
Antitumor efficacy-Duration of response (DOR) | 2 years
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause
Antitumor efficacy-Time to response (TTR) | 2 years
  Time from randomization to first recording of PR or CR

CONTACTS AND LOCATIONS:
Locations (1):
- Department of GI Oncology, Peking University Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No